CLINICAL TRIAL: NCT00750620
Title: A Phase 1, Open-Label, Single-Dose, Parallel-Group Study to Assess the Effect of Mild, Moderate and Severe Renal Impairment on the Pharmacokinetics of YM178
Brief Title: A Pharmacokinetic Study of YM178 in Normal Subjects and Those With Mild, Moderate, and Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 178-CL-038
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Renal Impairment
Keywords: mild, moderate, and severe renal impaired subjects; normal renal function subjects; Glomerular filtration rate (GFR); Modification of Diet in Renal Disease (MDRD) formula; YM178; pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency; Lymphoma, Follicular | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1. Severe renal impairment (Experimental): severe renal impairment
  Interventions: Drug: YM178
- 2. Moderate renal impairment (Experimental): moderate renal impairment
  Interventions: Drug: YM178
- 3. Mild renal impairment (Experimental): mild renal impairment
  Interventions: Drug: YM178
- 4. Normal renal function (Experimental): normal renal function
  Interventions: Drug: YM178

INTERVENTIONS:
Drug: YM178 — oral
  Other Names: mirabegron

SUMMARY:
The objective of this study is to assess and compare the pharmacokinetic properties of YM178 in normal subjects and those with mild, moderate and severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* good health other than renal impairment
* body mass index (BMI) between 18 and 40 kg/m2

Exclusion Criteria:

* subject with renal impairment has not been on stable dose of concomitant medication for at least 2 weeks
* subject has liver enzyme abnormalities

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetics parameters | day 1 - day 6

SECONDARY OUTCOMES:
Metabolite analysis | day 1 - day 6
Assessment of safety and tolerability | day 1 - day 6

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development
Locations (2):
- United States (2):
  - Anaheim, California
  - Miami, Florida

REFERENCES:
- [Background] Dickinson J, Lewand M, Sawamoto T, Krauwinkel W, Schaddelee M, Keirns J, Kerbusch V, Moy S, Meijer J, Kowalski D, Morton R, Lasseter K, Riff D, Kupcova V, van Gelderen M. Effect of renal or hepatic impairment on the pharmacokinetics of mirabegron. Clin Drug Investig. 2013 Jan;33(1):11-23. doi: 10.1007/s40261-012-0031-3. PMID 23208320